CLINICAL TRIAL: NCT06320158
Title: Dissecting the Molecular and Cellular Pathophysiology of Sarcopenic Obesity in the Elderly
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rovere Querini Patrizia, Principal Investigator, IRCCS San Raffaele
Other Study IDs: PNRR-MAD-2022-12376672
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenic Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who are candidates for hip surgery: cohort of patients who are candidates for hip surgery: completion of scales and questionnaires, venous blood sampling, muscle ultrasound scan
  Interventions: Other: clinical evaluation of sarcopenic obesity
- healthy subjects: cohort of healthy subjects recruited in 2016-2017 completion of scales, questionnaires and performance of the Short Physical Performance Battery test, venous blood sampling, muscle ultrasound scan
  Interventions: Other: clinical evaluation of sarcopenic obesity

INTERVENTIONS:
Other: clinical evaluation of sarcopenic obesity — completion of scales and questionnaires, venous blood sampling, muscle ultrasound scan

SUMMARY:
Ageing is characterised by a change in body composition with a parallel decrease in muscle mass and an increase and central redistribution of fat. When drastically exacerbated, these two processes culminate in a condition known as sarcopenic obesity (SO). SO is characterised by the coexistence of obesity and sarcopenia (i.e. reduced muscle mass and function) and is a growing public health problem in the elderly. The health risks of obesity and sarcopenia act synergistically, maximising the risk of disability of OS. The molecular mechanisms underlying OS are largely unknown. Increased fat mass induces chronic systemic inflammation and alters the profiles of adipokines and hormones, promoting the development of sarcopenia. On the other hand, the reduction in muscle tissue (SM) typical of sarcopenia is characterised by an alteration in the metabolic properties of skeletal muscle with an increase in insulin resistance and a reduction in energy expenditure that favours the accumulation and dysfunction of adipose tissue (AT). The cellular alterations that would seem to underlie OS are: altered autophagy, cellular senescence, epigenetic and mitochondrial alterations and maladaptive activation of intra- and intercellular inflammatory circuits (e.g. cytokines, extracellular vesicles, dysfunctional circulating leukocytes). However, the interconnections between these mechanisms are still unclear. The impact of OS can be dramatic on the health and quality of life of those affected. Therefore, the identification of early biomarkers that can recognise overweight and obese individuals at risk of developing SO is of paramount importance. This would shed light on the heterogeneity of an otherwise homogeneous clinical condition, opening new horizons towards the conscious design of more personalised therapeutic strategies, allowing a more rational use of the limited resources available for the growing elderly population.

The study design designed to achieve this aim is a cross-sectional observational study with an additional multicentre procedure lasting two years.

ELIGIBILITY:
Inclusion Criteria:

patients who are candidates for hip surgery

* patients who are candidates for hip surgery
* age ≥ 65 years
* patients able to give consent

healthy subjects

- healthy subjects from the geriatric cohort studied in 2016-2017 who at that time were: were overweight (25 ≤ BMI < 30 kg/m2) or obese (BMI ≥ 30 kg/m2) but had not yet developed sarcopenia

Exclusion Criteria:

All partecipants

* unavailability to participate in the study
* inflammatory or neurological myopathies
* acute heart failure
* active cancer

Ages: 65 Years to 99 Years | Sex: All
Age Groups: Older Adult
Study Population: patients who are candidates for hip surgery: 60 patients who are candidates for hip surgery. Specifically, we will select 15 obese and sarcopenic patients, 15 obese and non-sarcopenic patients, 15 non-obese and sarcopenic patients, and 15 non-obese and non-sarcopenic patients.
  healthy subjects:subjects from a previous cohort of healthy volunteers studied in 2016-2017. In particular, we will select overweight or obese subjects who did not have sarcopenia at the time of the 2016-2017 evaluation
Sampling Method: Non-Probability Sample
Enrollment: 1108 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identifying new molecular markers in elderly patients with sarcopenic obesity | May 2023- October 2024
  Identifying new molecular markers in elderly patients with sarcopenic obesity

SECONDARY OUTCOMES:
Assessing the ability of new markers (identified in the pre-clinical phase of this project) to predict individual disease trajectories | May 2023- October 2024
  Assessing the ability of new markers (identified in the pre-clinical phase of this project) to predict individual disease trajectories

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided